CLINICAL TRIAL: NCT00711516
Title: Double-Blind, Placebo-Controlled, Functional Neuroimaging Study of Armodafinil (200 mg/Day) on Prefrontal Cortical Activation in Patients With Residual Excessive Sleepiness Associated With Obstructive Sleep Apnea/Hypopnea
Brief Title: Study to Evaluate Armodafinil Treatment in Improving Prefrontal Cortical Activation and Working Memory Performance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C10953/4026/AP/US
Record Dates: First submitted 2008-07-08; First posted 2008-07-09 (Estimated); Results first posted 2011-02-14 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Excessive Sleepiness
MeSH Terms: conditions — Disorders of Excessive Somnolence | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Armodafinil treatment (200 mg/day) - Study drug was supplied as 50 mg tablets and the dose was titrated from a starting dose of 50 mg taken once daily in the morning (before 0800), increasing to 100 mg/day on Day 2, 150 mg/day on day 5, and then 200 mg/day beginning Day 8 and continuing through the end of the two week double-blind treatment period.
  Interventions: Drug: Armodafinil
- 2 (Placebo Comparator): Placebo comparator - Placebo tablets matching the armodafinil 50 mg tablets drug were supplied and the dose was titrated from a starting dose of one tablet taken once daily in the morning (before 0800), increasing to two tablets/day on Day 2, three tablets/day on day 5, and then four tablets/day beginning Day 8 and continuing through the end of the two week double-blind treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Armodafinil — Armodafinil once-daily (50 mg/day (1 tablet) on Day 1; increased to 100 mg/day (2 tablets) starting on Day 2; increased to 150 mg/day (3 tablets) starting on Day 5; increased to 200 mg/day (4 tablets) starting on Day 8). Then continue 200 mg/day dosage through Day 14.
  Arms: 1
Drug: Placebo — Matching Placebo dosed once-daily (50 mg/day (1 tablet) on Day 1; increased to 100 mg/day (2 tablets) starting on Day 2; increased to 150 mg/day (3 tablets) starting on Day 5; increased to 200 mg/day (4 tablets) starting on Day 8). Then continue 200 mg/day dosage through Day 14.
  Arms: 2

SUMMARY:
The primary objective of this study is to determine whether treatment with armodafinil will provide improvements in prefrontal cortical activation in patients with OSAHS (Obstructive Sleep Apnea/Hypopnea Syndrome) who have residual sleepiness despite receiving nCPAP therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a current diagnosis of OSAHS and has a complaint of excessive sleepiness despite effective nCPAP therapy.
* Patient has excessive sleepiness as evidenced by a mean sleep latency of less than 8 minutes, as determined by the MSLT.
* Patient has an ESS score of 10 or more at the initial screening visit.
* Patient has a habitual sleep time beginning no earlier than 2100 and ending no later than 0700.
* Patient is right-handed. Patients who are ambidextrous may be eligible following consultation with the medical monitor.
* Women of childbearing potential must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study.
* Patient exhibits reasonable accuracy (≥80%) on the 2-back working memory task during the training session at the second screening visit.

Exclusion Criteria:

The Patient:

* The patient is a current smoker or has a prior history of smoking (defined as ≥1 pack-year) within 2 years prior to the screening visit.
* consumes caffeine including coffee, tea and/or other caffeine-containing beverages or food averaging more than 400 mg of caffeine per day (approximately equivalent to 4 or more cups of coffee).
* has NART-predicted verbal IQ and QIDS-SR16 scores within protocol-specific exclusionary ranges.
* has a clinically significant, uncontrolled medical or psychiatric conditions (treated or untreated).
* has a confirmed or probable diagnosis of a current sleep disorder other than OSAHS.
* has used any excluded prescription drugs or procedures for prohibited and allowed drugs within the excluded timeframe.
* has a history of alcohol, narcotic, or any other drug abuse.
* has a positive UDS, without medical explanation, at the screening visit.
* has a clinically significant deviation from normal in the physical examination.
* is a pregnant or lactating woman. Any woman becoming pregnant during the study will be withdrawn from the study.
* has a past or present seizure disorder, head trauma that is clinically significant, or past neurosurgery.
* has used an investigational drug within 1 month before the screening visit.
* has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery).
* has a known hypersensitivity to armodafinil or modafinil, or any other component of the study drug tablets.
* has a history of any clinically significant cutaneous drug reaction, or a history of clinically significant hypersensitivity reaction, including multiple allergies or drug reactions.
* has known human immunodeficiency virus (HIV).
* has clinical laboratory test value(s) outside the range(s) specified in the Protocol, or presents a clinically significant laboratory abnormality without prior written approval by the medical monitor.
* has worked the night shift within 28 days of the baseline visit, or will work the night shift during the double-blind segment of the study.
* anticipates any travel across more than 3 time zones at any time during the study.
* needs to use any of the excluded medications identified in this protocol.
* is unable to complete neuroimaging studies, performance tasks, self-rating scales, and all other study assessments.
* has a contraindication to fMRI scanning, (such as an implanted pacemaker/defibrillator, aneurysm clips, drug infusion device or metallic foreign body).
* is suspected to be unable to tolerate fMRI scanning (eg, claustrophobic) and/or the testing paradigm.
* has physical or other characteristics that suggest imaging data will be unobtainable or degraded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (9):
- United States (9):
  - Peninsula Sleep Center, Burlingame, California
  - Pacific Research, San Diego, California
  - VA San Diego Healthcare System, San Diego, California
  - Stanford University, Stanford, California
  - Beth Israel Deaconess Medical, Boston, Massachusetts
  - Neurocare, Inc., Newton, Massachusetts
  - Washington University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Wake Research Associates, Raleigh, North Carolina

REFERENCES:
- [Derived] Greve DN, Duntley SP, Larson-Prior L, Krystal AD, Diaz MT, Drummond SP, Thein SG, Kushida CA, Yang R, Thomas RJ. Effect of armodafinil on cortical activity and working memory in patients with residual excessive sleepiness associated with CPAP-Treated OSA: a multicenter fMRI study. J Clin Sleep Med. 2014 Feb 15;10(2):143-53. doi: 10.5664/jcsm.3440. PMID 24532997

RESULTS

PARTICIPANT FLOW:
Groups:
- Armodafinil (200 mg/Day): Armodafinil was titrated during the double-blind treatment period starting with 50 mg/day (1 tablet) on Day 1, increasing to 100 mg/day (2 tablets) on day 2, 150 mg/day (3 tablets) on day 5, and 200 mg/day (4 tablets) on day 8, which was continued for the remainder of the 2-week double-blind treatment period.
- Placebo: Placebo tablets matching the armodafinil tablets were titrated during the double-blind treatment period starting with 1 tablet/day on Day 1, increasing to 2 tablets/day on day 2, 3 tablets/day on day 5, and 4 tablets/day on day 8, which was continued for the remainder of the 2-week double-blind treatment period.
Period: Overall Study
Arm/Group | Armodafinil (200 mg/Day) | Placebo
Started | 21 | 19
Completed | 20 | 16
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armodafinil (200 mg/Day) | Placebo | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 19 | 40
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49.9 (8.98) | 50.7 (7.95) | 50.3 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 17 | 14 | 31
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint in Number of Contiguous Activated Voxels Meeting Predefined Threshold in Dorsolateral Prefrontal Cortex (DLPFC) on Functional Magnetic Resonance Imaging (fMRI) as a Measure of Prefrontal Cortical Activation
Description: The primary outcome was the change from baseline in number of contiguous activated voxels in the dorsolateral prefrontal cortex (DLPFC) on functional magnetic resonance imaging (fMRI) at Week 2(or last observation after baseline). Each voxel is compared to the reference wave form. If it differs from that value p<0.05, the voxel is considered active. fMRI is a brain imaging technique that identifies neuronal activation related to specific tasks or sensory stimulation. Increased neuronal activity increases blood flow and oxygen content to the activated part of the brain, altering fMRI signal.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Efficacy analyses were performed on the full analysis dataset which includes those patients in the safety analysis set who had at least 1 post baseline primary efficacy assessment.
Measure: Mean (Standard Deviation); unit: Activated voxels
Groups:
- Armodafinil: Armodafinil was provided to patients in bottles of sixty 50 mg tablets. Patients took a 50 mg dose on Day 1, which was increased by 50 mg on Days 2, 5, and 8 to a total dose of 200 mg per day. This was taken as a once daily dose at or before 8 AM, approximately 30 minutes before breakfast.
- Placebo: Placebo tablets matching the 50 mg armodafinil tablets were provided by Cephalon to patients in bottles of sixty tablets. Patients took a single tablet on Day 1, which was increased by 1 tablet on Days 2, 5, and 8 to a total dose of 4 tablets per day. This was taken as a once daily dose at or before 8 AM, approximately 30 minutes before breakfast.
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Activated voxels | -1932.3 (2993.8) | -2428.1 (5023.53)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Using the standardized difference of 1.10, 28 evaluable patients (14 per treatment group) were required to provide 80% power while controlling the 2-sided, Type 1 error rate at 0.05. With an estimated 25% attrition rate, a total of 38 patients (19 per group) were planned. First analyzed using ANCOVA,the residuals were used to test for normality using Shapiro-Wilk; normality was violated therefore treatment comparison used the Wilcoxon rank sum; Test type: Superiority or Other; p = 0.7382, Wilcoxon (Mann-Whitney) — The hierarchical testing procedure was employed to control the studywise error rate at 0.05; The assumption of normality was violated (p-value ≤0.05), therefore the treatment comparison was made using a Wilcoxon rank-sum test; Median Difference (Net) = -241.8, 95% CI 2-sided [-2470.0 to 2102.3]

2. Secondary Outcome: Change From Baseline to Endpoint in Mean Response Latency in the 2-Back Working Memory Test at Endpoint - Mean Performance Speed
Description: The 2-Back is a verbal working memory test in which random letters are presented visually every 4 sec, with each stimulus lasting 500 msec. Subjects are asked to make a yes/no response following each letter indicating whether it was the same or different from the letter presented two earlier. The load on working memory was the ordering, retention, updating, and manipulation of 2 letters and consideration of the relationship to a 3rd newly presented letter, which could have been a target or a nontarget. The change from baseline in response latency at endpoint is presented here.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy assessment after baseline.
Measure: Mean (Standard Deviation); unit: Milliseconds (ms)
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Milliseconds (ms) | 2.3 (78.94) [-171.9 to 181.3] | -59.0 (112.69) [-258.4 to 89.1]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; The statistical hypothesis for this key secondary efficacy variable was to be tested using the same model as specified for the primary objective efficacy variable (ANCOVA, ANOVA, and Wilcoxon as appropriate). All statistical tests were 2 tailed at the 0.05 level of significance; Test type: Superiority or Other; p = 0.1661, Wilcoxon (Mann-Whitney); Median Difference (Net) = 53.2, 95% CI 2-sided [-17.8 to 136.1]

3. Secondary Outcome: Change From Baseline to Endpoint in the Number of Contiguous Activated Voxels Meeting the Predefined Threshold in the Anterior Cingulate Cortex (ACC)
Description: The outcome was the change from baseline in number of contiguous activated voxels in the anterior cingulate cortex (ACC) on functional magnetic resonance imaging (fMRI) at Week 2(or last observation after baseline). Each voxel is compared to the reference wave form. If it differs from that value p<0.05, the voxel is considered active. fMRI is a brain imaging technique that identifies neuronal activation related to specific tasks or sensory stimulation. Increased neuronal activity increases blood flow and oxygen content to the activated part of the brain, altering fMRI signal.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy assessment after baseline
Measure: Mean (Standard Deviation); unit: Activated Voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Activated Voxels | -107.3 (367.92) | -206.5 (340.56)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.5774, Wilcoxon (Mann-Whitney); Median Difference (Net) = 78.9, 95% CI 2-sided [-157.8 to 311.3]

4. Secondary Outcome: Change From Baseline to Endpoint in the Number of Contiguous Voxels Meeting the Predefined Threshold in the Posterior Parietal Cortex (PPC)
Description: The outcome was the change from baseline in number of contiguous activated voxels in the posterior parietal cortex (PPC) on functional magnetic resonance imaging (fMRI) at Week 2(or last observation after baseline). Each voxel is compared to the reference wave form. If it differs from that value with p<0.05, the voxel is considered active. fMRI is a brain imaging technique that identifies neuronal activation related to specific tasks or sensory stimulation. Increased neuronal activity increases blood flow and oxygen content to the activated part of the brain, altering fMRI signal.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy assessment after baseline
Measure: Mean (Standard Deviation); unit: Activated voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Activated voxels | -595.0 (1251.79) | -773.3 (1693.48)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.8610, Wilcoxon (Mann-Whitney); Median Difference (Net) = 90.1, 95% CI 2-sided [-806.7 to 707.0]

5. Secondary Outcome: Change From Baseline to Endpoint in the Number of Contiguous Activated Voxels Meeting the Predefined Threshold in the Thalamus
Description: The outcome was the change from baseline in number of contiguous activated voxels in the thalamus on functional magnetic resonance imaging (fMRI) at Week 2(or last observation after baseline). Each voxel is compared to the reference wave form. If it differs from that value significantly (p<0.05), the voxel is considered active. fMRI is a brain imaging technique that identifies neuronal activation related to specific tasks or sensory stimulation. Increased neuronal activity increases blood flow and oxygen content to the activated part of the brain, altering fMRI signal.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: Activated voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Activated voxels | -841.7 (401.77) | -1417.9 (638.48)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.6907, Wilcoxon (Mann-Whitney); Median Difference (Net) = 252.8, 95% CI 2-sided [-1066.5 to 1523.8]

6. Secondary Outcome: Pattern Recognition Memory (PRM) Percent Correct (Immediate) From the CANTAB Battery-Change From Baseline to Endpoint
Description: The PRM test from the Cambridge Neuropsychological Test Automated Battery (CANTAB) assesses episodic memory by a patient's ability to encode and recognize visual information. Patterns appear sequentially on the screen, and patients are instructed to remember them. Immediately afterwards a recognition test is performed, in which each pattern shown earlier is presented with another pattern of similar form and color. Patient has to touch the pattern seen earlier. Change from baseline to endpoint in % correct responses with immediate recall is presented. Subjects complete 24 trials per assessment.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy evaluation after baseline
Measure: Mean (Standard Deviation); unit: Percent correct trials
Units Other Than Participants: trials
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Number analyzed (trials) | 24 | 24
Percent correct trials | -0.1 (6.56) | 3.2 (6.77)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.2456, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0.0, 95% CI 2-sided [-8.0 to 0.0]

7. Secondary Outcome: Pattern Recognition Memory (PRM) Percent Correct (Delayed) From the CANTAB Battery-Change From Baseline to Endpoint
Description: The PRM test from the Cambridge Neuropsychological Test Automated Battery (CANTAB) assesses episodic memory as measured by a patient's ability to encode and recognize visual information. Patterns appear sequentially on the screen, and patients are instructed to remember them. Twenty minutes following the immediate recognition test, another "delayed" recognition test is performed, featuring the same stimuli as in the first phase. The change from baseline to endpoint in percent correct responses of this delayed test are presented here. Subjects complete 24 trials per assessment.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy evaluation after baseline
Measure: Mean (Standard Deviation); unit: Percent correct trials
Units Other Than Participants: Trials
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 19 | 16
Number analyzed (Trials) | 24 | 24
Percent correct trials | 0.4 (12.34) | -1.1 (10.70)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.7115, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0, 95% CI 2-sided [-8.0 to 9.0]

8. Secondary Outcome: Reaction Time Index (RTI) Median Correct Latency, Five Choice Test From the CANTAB Battery-Change From Baseline to Endpoint
Description: The RTI is a measure of simple and choice reaction time, movement time and spatio-temporal vigilance during simple and 5 choice reaction time trials. This task also permits measurement of anticipatory/premature responding and perseverative responding. The patient responded to a yellow spot appearing on the screen by letting go of the press pad and touching the location in which the spot appeared. The yellow spot appeared in any 1 of 5 locations in the 5 choice reaction time phase. The change from baseline to endpoint in median correct latency is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy assessment after baseline
Measure: Median (Full Range); unit: Milliseconds (ms)
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Milliseconds (ms) | -6.5 [-54.0 to 47.0] | -12.5 [-252.0 to 44.0]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.6103, Wilcoxon (Mann-Whitney); Median Difference (Net) = 4.0, 95% CI 2-sided [-13.0 to 19.0]

9. Secondary Outcome: Reaction Time Index (RTI) Median Correct Latency, One Choice Test From the CANTAB Battery-Change From Baseline to Endpoint
Description: The RTI is a measure of simple and choice reaction time, movement time and spatio-temporal vigilance during simple and 5 choice reaction time trials. This task also permits measurement of anticipatory/premature responding and perseverative responding. The patient responded to a yellow spot appearing on the screen by letting go of the press pad and touching the location in which the spot appeared. The yellow spot appeared in a single location during the simple reaction time phase. The change from baseline to endpoint in median correct latency is presented here.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy assessment after baseline
Measure: Median (Full Range); unit: Milliseconds (ms)
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Milliseconds (ms) | -13.5 [-45.0 to 37.0] | -4.5 [-224.0 to 39.0]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.9619, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0.0, 95% CI 2-sided [-18.0 to 17.0]

10. Secondary Outcome: One Touch Stockings of Cambridge (OTS) Mean Correct Latency, (Easy) From the CANTAB Battery-Change From Baseline to Endpoint
Description: OTS is a spatial planning test based on Tower of London test and the CANTAB Stockings of Cambridge test, and measures frontal lobe function. Subject is shown 2 displays containing 3 colored balls and a row of boxes containing numbers. The patient was shown one demonstration problem and then had to solve 3 additional problems (easy). The problems increased in complexity, from one to six moves. With additional problems subject had to work out how many moves the solutions required in their heads (hard). Change from baseline to endpoint in Mean correct latency for the easy problems is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy assessment after baseline.
Measure: Mean (Standard Deviation); unit: Milliseconds (ms)
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Milliseconds (ms) | -787.9 (1198.06) | -666.7 (1751.66)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.4544, Wilcoxon (Mann-Whitney); Median Difference (Net) = -335.5, 95% CI 2-sided [-1270.7 to 723.3]

11. Secondary Outcome: One Touch Stockings of Cambridge (OTS) Mean Correct Latency, (Hard) From the CANTAB Battery-Change From Baseline to Endpoint
Description: OTS is a spatial planning test based on Tower of London test and the CANTAB Stockings of Cambridge test, and measures frontal lobe function. Subject is shown 2 displays containing 3 colored balls and a row of boxes containing numbers. The patient was shown one demonstration problem and then had to solve 3 additional problems (easy). The problems increased in complexity, from one to six moves. With additional problems subject had to work out how many moves the solutions required in their heads (hard). Change from baseline to endpoint in Mean correct latency for the hard problems is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy assessment after baseline
Measure: Mean (Standard Deviation); unit: Milliseconds (ms)
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Milliseconds (ms) | -733.3 (8352.4) | -6898.1 (8708.46)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.0193, Wilcoxon (Mann-Whitney); Median Difference (Net) = 6410.3, 95% CI 2-sided [1064.7 to 12087.3]

12. Secondary Outcome: One Touch Stockings of Cambridge (OTS) Mean Choices to Correct, (Easy) From the CANTAB Battery-Change From Baseline to Endpoint
Description: OTS is a spatial planning test based on the Tower of London and the CANTAB Stockings of Cambridge test, and measures frontal lobe function. Patient shown 2 displays containing 3 colored balls and a row of boxes containing numbers. The patient is shown one demonstration problem and then solves 3 additional problems (easy). Problems increased in complexity, from one to six moves. With additional problems (hard) the patient has to work out how many moves the solutions required in their heads. Mean change from Baseline to endpoint in number of choices to correct for easy problems is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy measure after baseline
Measure: Mean (Standard Deviation); unit: Choices to correct
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Choices to correct | 0.0 (0.08) | 0.0 (0.17)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.1704, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0.0, 95% CI 2-sided [-0.1 to 0.0]

13. Secondary Outcome: One Touch Stockings of Cambridge (OTS) Mean Choices to Correct, (Hard) From the CANTAB Battery-Change From Baseline to Endpoint
Description: OTS is a spatial planning test based on the Tower of London and the CANTAB Stockings of Cambridge test, and measures frontal lobe function. Patient shown 2 displays containing 3 colored balls and a row of boxes containing numbers. The patient was shown one demonstration problem and then solves 3 additional problems (easy). Problems increased in complexity, from one to six moves. With additional problems (hard) the patient had to work out how many moves the solutions required in their heads. Mean change from baseline to endpoint in number of choices to correct for hard problems is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy assessment after baseline
Measure: Mean (Standard Deviation); unit: Choices to correct
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Choices to correct | -0.2 (0.29) | 0.0 (0.30)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.0609, Wilcoxon (Mann-Whitney); Median Difference (Net) = -0.2, 95% CI 2-sided [-0.3 to 0.0]

14. Secondary Outcome: Epworth Sleepiness Scale Change From Baseline to Endpoint
Description: The patient's evaluation of excessive daytime sleepiness was measured by the patient reported measure, ESS (Johns1991). The ESS score was based on responses to questions referring to 8 everyday situations (eg, sitting and reading, talking to someone, being stopped in traffic) and reflected a patient's propensity to fall asleep in those situations. The ESS score was derived from the sum of the values from questions corresponding to the 8 situations. Scores for the ESS ranged from 0 to 24, with a higher score indicating a greater daytime sleepiness. Change from baseline to endpoint is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full analysis set defined as subjects who had at least one efficacy evaluation after baseline
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Units on a scale | -5.8 (1.03) | -2.9 (1.08)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Hierarchical testing procedure was used to control the studywise error rate at 0.05. If treatment was statistically significant on the primary variable, the key secondary variable would be claimed as significant if p-value was <= 0.05. If primary and key secondary variables were significant subsequent secondary variables following the order presented here would be claimed as significant if their p-values were <= 0.05. If any were >0.05 subsequent p-values would be reported as nominal p-values; Test type: Superiority or Other; p = 0.0499, ANCOVA — Nominal P-value for treatment comparison is from an analysis of covariance (ANCOVA) with treatment and center as factors and the baseline value as covariate; Mean Difference (Net) = -2.9, 95% CI 2-sided [-5.8 to -0.0]

15. Secondary Outcome: Clinical Global Impression of Change (CGI-C)- Number of Responders at Endpoint
Description: Severity of sleepiness, was assessed by the Clinical Global Impression of Severity (CGI-S) at Baseline. The clinician assessed the change from baseline in the patient's condition, as related to excessive sleepiness, in response to treatment using the CGI-C, which consisted of the following 7 categories and scoring assignments: very much improved, much improved, minimally improved, no change, minimally worse, much worse, and very much worse. Responders had to be at least minimally improved from Baseline to qualify as a responder at Endpoint.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy assessment after baseline
Measure: Number; unit: Participants
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Participants | 13 | 9
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.7343, Fisher Exact

16. Secondary Outcome: Total Score From the Medical Outcomes Study 6-Item Cognitive Function Scale (MOS-CF6)-Change From Baseline to Endpoint
Description: The MOS-CF6 is an instrument to assess patient self-reported cognitive function. Items were selected to cover 6 relevant aspects of cognitive functioning as follows: confusion, concentration/thinking, attention, memory, reasoning, problem solving, and processing speed. The CF 6 item responses include 6 choices, ranging from "none of the time" to "all of the time." The CF-6 was scored by summing responses across the 6 items and converting the total to a 0 to 100 point scale, with higher scores indicating better cognitive functioning. Change in MOS-CF6 from baseline to endpoint is reported.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Population defined as subjects who had at least one efficacy evaluation after baseline.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Units on a scale | 6.1 (2.82) | -0.2 (3.11)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.1246, ANCOVA — P-value for the treatment comparison is from an analysis of covariance (ANCOVA) with treatment and center as factors and the baseline value as a covariate; Mean Difference (Net) = 6.2, 95% CI 2-sided [-1.8 to 14.3]

17. Secondary Outcome: Blood Oxygenation Level Dependent (BOLD) Signal Intensity - Percent Change From Baseline to Endpoint in the Dorsolateral Prefrontal Cortex (DLPFC)
Description: Functional magnetic resonance imaging (fMRI) is a brain imaging technique that identifies neuronal activation in regions related to specific tasks or sensory stimulation such as language, vision, hearing, and short-term memory. When neuronal activity increases, blood flow increases to that part of the brain with an increase in the oxygen content of the blood. Increase in oxygen content causes the fMRI signal in that part of the brain to change, and is the basis of the BOLD effect. The percent change in BOLD signal from Baseline to 2 weeks or last observation after baseline is presented here.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy assessment after baseline.
Measure: Median (Full Range); unit: Percentage change in BOLD signal
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Percentage change in BOLD signal | -0.398 (4.2761) [-23.439 to 45.139] | 4.704 (10.3232) [-43.840 to 94.919]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.7382, Wilcoxon (Mann-Whitney); Median Difference (Net) = -4.026, 95% CI 2-sided [-21.684 to 19.980]

18. Secondary Outcome: Blood Oxygenation Level Dependent (BOLD) Signal Intensity - Percent Change From Baseline to Endpoint in the Anterior Cingulate Cortex (ACC)
Description: as for outcome 17
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects with at least one efficacy evaluation after baseline
Measure: Median (Full Range); unit: Percent change in BOLD signal
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Percent change in BOLD signal | -1.777 (6.7798) [-38.587 to 99.034] | 7.148 (9.4912) [-100.0 to 55.958]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 1.000, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0.086, 95% CI 2-sided [-19.195 to 25.043]

19. Secondary Outcome: Blood Oxygenation Level Dependent (BOLD) Signal Intensity -Change From Baseline to Endpoint in the Posterior Parietal Cortex (PPC)
Description: as for outcome 17
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy evaluation after baseline
Measure: Median (Full Range); unit: Percent change in Bold signal
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Percent change in Bold signal | 3.199 (3.2493) [-31.541 to 27.343] | -2.021 (4.9907) [-30.116 to 32.956]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.8861, Wilcoxon (Mann-Whitney); Median Difference (Net) = 1.282, 95% CI 2-sided [-11.460 to 14.770]

20. Secondary Outcome: Blood Oxygenation Level Dependent (BOLD) Signal Intensity - Percent Change From Baseline to Endpoint in the Thalamus
Description: as for outcome 17
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one efficacy evaluation after baseline
Measure: Median (Full Range); unit: Percent change in BOLD signal
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Percent change in BOLD signal | 16.363 (9.6289) [-41.089 to 98.265] | 2.099 (7.7566) [-30.301 to 74.962]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.4738, Wilcoxon (Mann-Whitney); Median Difference (Net) = 11.825, 95% CI 2-sided [-12.601 to 37.987]

21. Secondary Outcome: Activation-Performance Relationship Between the Functional Magnetic Resonance Imaging (fMRI) in Dorsolateral Prefrontal Cortex (DLPFC) and 2-Back Working Memory Test - Number of Voxels Activated at Endpoint
Description: With this outcome measure the correlation between the number of voxels activated on fMRI (voxels that differ significantly from reference wave form) in DLPFC versus performance on the 2-back working memory test was evaluated for both Armodafinil and Placebo. Correlation coefficients and P-values are presented for each treatment group.
Time Frame: Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects with at least one observation after baseline
Measure: Number; unit: Correlation Coefficient
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Correlation Coefficient | 0.422 [-0.026 to 0.728] | -0.445 [-0.770 to 0.066]
Statistical Analysis 1: Comparison: Armodafinil; Pearson's correlation coefficient was used to assess the relationship between fMRI variable and performance on the 2-back working memory test; Test type: Superiority or Other; p = 0.0573, Pearson's Correlation Coefficient; The SAS CORR procedure was used to analyze the activation performance relationships. All estimations are based on Fisher's z-transformation
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p = .0754, Pearson's Correlation Coefficient; [statistical method as in outcome 21, analysis 1]

22. Secondary Outcome: Activation-Performance Relationship Between the Functional Magnetic Resonance Imaging (fMRI) in Anterior Cingulate Cortex (ACC) and 2-Back Working Memory Test - Number of Voxels Activated at Endpoint
Description: With this outcome measure the correlation between the number of voxels activated on fMRI (voxels that differ significantly from reference wave form) in ACC versus performance on the 2-back working memory test was evaluated for both Armodafinil and Placebo. Correlation coefficients and P-values are presented for each treatment group.
Time Frame: Week 2 or Last Observation after Baseline
Population: Full Analysis Set defined as subjects with at least one efficacy evaluation after baseline
Measure: Number; unit: Correlation Coefficient
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Correlation Coefficient | 0.254 [-0.213 to 0.626] | -0.152 [-0.603 to 0.371]
Statistical Analysis 1: Comparison: Armodafinil; Test type: Superiority or Other; p = 0.2727, Pearson's Correlation Coefficient
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p = .5671, Pearson's Correlation Coefficient

23. Secondary Outcome: Activation-Performance Relationship Between Functional Magnetic Resonance Imaging (fMRI) in Posterior Parietal Cortex (PPC) and the 2-Back Working Memory Test -Number of Voxels Activated at Endpoint
Description: With this outcome measure the correlation between the number of voxels activated on fMRI (voxels that differ significantly from reference wave form) in PPC versus performance on the 2-back working memory test was evaluated for both Armodafinil and Placebo. Correlation coefficients and P-values are presented for each treatment group.
Time Frame: Week 2 or Last Observation after Baseline
Population: Full Analysis Set defined as subjects with at least one observation after baseline
Measure: Number; unit: Correlation Coefficient
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Correlation Coefficient | 0.355 [-0.104 to 0.689] | -0.358 [-0.725 to 0.168]
Statistical Analysis 1: Comparison: Armodafinil; Test type: Superiority or Other; p = 0.1169, Pearson's Correlation Coefficient; [statistical method as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p = 0.1634, Pearson's Correlation Coefficient; [statistical method as in outcome 21, analysis 1]

24. Secondary Outcome: Activation-Performance Relationship Between Functional Magnetic Resonance Imaging (fMRI) in the Thalamus and 2-Back Working Memory Test -Number of Voxels Activated at Endpoint
Description: With this outcome measure the correlation between the number of voxels activated on fMRI (voxels that differ significantly from reference wave form) in the thalamus versus performance on the 2-back working memory test was evaluated for both Armodafinil and Placebo. Correlation coefficients and P-values are presented for each treatment group.
Time Frame: Week 2 or Last Observation after Baseline
Population: Full Analysis Set defined as subjects with at least one observation after baseline
Measure: Number; unit: Correlation Coefficient
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Correlation Coefficient | 0.405 [-0.046 to 0.719] | -0.038 [-0.524 to 0.467]
Statistical Analysis 1: Comparison: Armodafinil; Test type: Superiority or Other; p = 0.0692, Pearson's Correlation Coefficient; [statistical method as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p = .8876, Pearson's Correlation Coefficient; [statistical method as in outcome 21, analysis 1]

25. Secondary Outcome: Activation-Performance Relationship Between the Functional Magnetic Resonance Imaging (fMRI) in Dorsolateral Prefrontal Cortex (DLPFC) and 2-Back Working Memory Test - Blood Oxygen Level Dependent (BOLD) Signal Intensity at Endpoint
Description: With this outcome measure the correlation between the BOLD signal intensity on fMRI over DLPFC versus performance on the 2-back working memory test was evaluated for both Armodafinil and Placebo. Correlation coefficients and P-values are presented for each treatment group.
Time Frame: Week 2 or Last Observation after Baseline
Population: Full Analysis Set defined as subjects with at least one observation after baseline
Measure: Number; unit: Correlation Coefficient
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Correlation Coefficient | -0.122 [-0.536 to 0.339] | 0.789 [0.481 to 0.923]
Statistical Analysis 1: Comparison: Armodafinil; Test type: Superiority or Other; p = 0.6030, Pearson's Correlation Coefficient; [statistical method as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p < .0001, Pearson's Correlation Coefficient; [statistical method as in outcome 21, analysis 1]

26. Secondary Outcome: Activation-Performance Relationship Between Functional Magnetic Resonance Imaging (fMRI) in Anterior Cingulate Cortex (ACC) and 2-Back Working Memory Test -Blood Oxygen Level Dependent (BOLD) Signal Intensity at Endpoint
Description: With this outcome measure the correlation between the BOLD signal intensity on fMRI in the ACC versus performance on the 2-back working memory test was evaluated for both Armodafinil and Placebo. Correlation coefficients and P-values are presented for each treatment group.
Time Frame: Week 2 or Last Observation after Baseline
Population: Full Analysis Set defined as subjects with at least one observation after baseline
Measure: Number; unit: Correlation Coefficient
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Correlation Coefficient | 0.025 [-0.423 to 0.462] | -0.012 [-0.505 to 0.487]
Statistical Analysis 1: Comparison: Armodafinil; Test type: Superiority or Other; p = 0.9170, Pearson's Correlation Coefficient; [statistical method as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p = .9642, Pearson's Correlation Coefficient; [statistical method as in outcome 21, analysis 1]

27. Secondary Outcome: Activation-Performance Relationship on Functional Magnetic Resonance Imaging (fMRI) in Posterior Parietal Cortex (PPC) and 2-Back Working Memory Test - Blood Oxygen Level Dependent (BOLD) Signal Intensity at Endpoint
Description: With this outcome measure the correlation between the BOLD signal intensity on fMRI in PPC versus performance on the 2-back working memory test was evaluated for both Armodafinil and Placebo. Correlation coefficients and P-values are presented for each treatment group.
Time Frame: Week 2 or Last Observation after Baseline
Population: Full Analysis Set defined as subjects with at least one observation after baseline
Measure: Number; unit: Correlation Coefficient
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Correlation Coefficient | 0.065 [-0.388 to 0.494] | 0.364 [-0.161 to 0.728]
Statistical Analysis 1: Comparison: Armodafinil; Test type: Superiority or Other; p = 0.7813, Pearson's Correlation Coefficient; [statistical method as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p = 0.1560, Pearson's Correlation Coefficient; [statistical method as in outcome 21, analysis 1]

28. Secondary Outcome: Activation-Performance Relationship on Functional Magnetic Resonance Imaging (fMRI) in the Thalamus and 2-Back Working Memory Test - Blood Oxygen Level Dependent (BOLD) Signal Intensity at Endpoint
Description: With this outcome measure the correlation between BOLD signal intensity on fMRI in the thalamus versus performance on the 2-back working memory test was evaluated for both Armodafinil and Placebo. Correlation coefficients and P-values are presented for each treatment group.
Time Frame: Week 2 or Last Observation after Baseline
Population: Full Analysis Set defined as subjects with at least one observation after baseline
Measure: Number; unit: Correlation Coefficient
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 20 | 16
Correlation Coefficient | -0.029 [-0.466 to 0.419] | 0.582 [0.121 to 0.836]
Statistical Analysis 1: Comparison: Armodafinil; Test type: Superiority or Other; p = 0.9010, Pearson's Correlation Coefficient; [statistical method as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p = 0.0135, Pearson's Correlation Coefficient; [statistical method as in outcome 21, analysis 1]

29. Secondary Outcome: Number of Contiguous Activated Voxels Meeting Predefined Threshold in the DLPFC on fMRI on the 2 Back Working Memory Test - Change From Baseline-Subgroup-Responders in 2 Back Working Memory Test
Description: This is a subgroup analysis of responders on the 2-back working memory test for the number of voxels meeting the predefined threshold in DLPFC. A responder in the 2-back working memory test was defined as a patient showing a response latency of less than 713 ms at endpoint. This is based on baseline data from the matched control population in a functional imaging study in patients with obstructive sleep apnea. The change from Baseline to Endpoint in the number of activated voxels (that differ significantly from reference wave form) for each treatment group among the responders is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Sub-group Analysis of subjects who were responders on the 2-Back Working Memory Test defined as subjects who had a response latency of < 713 ms at Endpoint
Measure: Mean (Standard Error); unit: Activated voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 8 | 4
Activated voxels | -1411.6 (1365.62) | -1359.0 (1146.49)

30. Secondary Outcome: Number of Contiguous Activated Voxels Meeting Predefined Threshold in the ACC on fMRI by 2-Back Working Memory Test -Change From Baseline; Subgroup-Responders in 2 Back Memory Test
Description: This is a subgroup analysis of responders on the 2-back working memory test for the number of activated voxels (that differ significantly from reference wave form) in Anterior Cingulate Cortex (ACC). A responder in the 2-back working memory test was defined as a patient showing a response latency of less than 713 ms at endpoint. This is based on baseline data from the matched control population in a functional imaging study in patients with obstructive sleep apnea. The change from Baseline to Endpoint in the number of activated voxels for each treatment group among the responders is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Sub-group Analysis of subjects who were responders on the 2-Back Working Memory Test (had response latency < 713 ms) at Endpoint
Measure: Mean (Standard Error); unit: Voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 8 | 4
Voxels | -38.6 (113.68) | -227.8 (213.46)

31. Secondary Outcome: Number of Contiguous Activated Voxels Meeting Predefined Threshold in the PPC on fMRI by 2-Back Working Memory Test-Change From Baseline; Subgroup-Responders in 2 Back Memory Test
Description: This is a subgroup analysis of responders on the 2-back working memory test for the number of voxels (voxels that differ significantly from reference wave form) in Posterior Parietal Cortex (PPC). A responder in the 2-back working memory test was defined as a patient showing a response latency of less than 713 ms at endpoint. This is based on baseline data from the matched control population in a functional imaging study in patients with obstructive sleep apnea. The change from Baseline to Endpoint in the number of activated voxels for each treatment group among the responders is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Sub-group Analysis of subjects who were responders on the 2-Back Working Memory Test (had a response latency < 713 ms) at Endpoint
Measure: Mean (Standard Error); unit: Voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 8 | 4
Voxels | -789.1 (588.22) | -397.7 (366.33)

32. Secondary Outcome: Number of Contiguous Activated Voxels Meeting Predefined Threshold in the Thalamus on fMRI by 2-Back Working Memory Test-Change From Baseline; Subgroup-Responders in 2 Back Memory Test
Description: This is a subgroup analysis of responders on the 2-back working memory test for the number of activated voxels (voxels that differ significantly from reference wave form) in the thalamus. A responder in the 2-back working memory test was defined as a patient showing a response latency of less than 713 ms at endpoint. This is based on baseline data from the matched control population in a functional imaging study in patients with obstructive sleep apnea. The change from Baseline to Endpoint in the number of activated voxels for each treatment group among the responders is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Sub-group Analysis of subjects who were responders on the 2-Back Working Memory Test (response latency < 713 ms) at Endpoint
Measure: Mean (Standard Error); unit: Voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 8 | 4
Voxels | -764.7 (626.55) | -1446.7 (1091.13)

33. Secondary Outcome: Number of Contiguous Activated Voxels Meeting Predefined Threshold in the DLPFC on fMRI by 2-Back Working Memory Test-Change From Baseline; Subgroup-Non Responders in 2 Back Memory Test
Description: This is a subgroup analysis of non-responders on the 2-back working memory test for the number of voxels meeting the predefined threshold (voxels that differ significantly from reference wave form) on functional magnetic resonance imaging (fMRI). A non-responder in the 2-back working memory test was defined as a patient showing a response latency of 713 ms or greater at endpoint. The change from Baseline to Endpoint in the number of activated voxels in the dorsolateral prefrontal cortex (DLPFC)for each treatment group among the non-responders is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Sub-group analysis among non-responders on the 2-Back Working Memory Test (response latency of 713 ms or greater) at Endpoint
Measure: Mean (Standard Error); unit: Voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 12 | 12
Voxels | -2279.4 (686.69) | -2784.4 (1643.79)

34. Secondary Outcome: Number of Contiguous Activated Voxels Meeting Predefined Threshold in the ACC on fMRI by 2-Back Working Memory Test-Change From Baseline; Subgroup-Non Responders in 2 Back Memory Test
Description: This is a subgroup analysis of non-responders on the 2-back working memory test for the number of voxels meeting the predefined threshold (voxels that differ significantly from reference wave form) on functional magnetic resonance imaging (fMRI). A non-responder in the 2-back working memory test was defined as a patient showing a response latency of 713 ms or greater at endpoint. The change from Baseline to Endpoint in the number of activated voxels in the anterior cingulate cortex (ACC)for each treatment group among the non-responders is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Sub-group analysis of non-responders on the 2-Back Working Memory Test (response latency of 713 ms or greater) at Endpoint
Measure: Mean (Standard Error); unit: Voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 12 | 12
Voxels | -153.1 (116.30) | -199.4 (94.97)

35. Secondary Outcome: Number of Contiguous Activated Voxels Meeting Predefined Threshold in the PPC on fMRI by 2-Back Working Memory Test-Change From Baseline; Subgroup-Non Responders in 2 Back Memory Test
Description: This is a subgroup analysis of non-responders on the 2-back working memory test for the number of voxels meeting the predefined threshold (voxels that differ significantly from reference wave form) on functional magnetic resonance imaging (fMRI). A non-responder in the 2-back working memory test was defined as a patient showing a response latency of 713 ms or greater at endpoint. The change from Baseline to Endpoint in the number of activated voxels in the posterior parietal cortex (PPC)for each treatment group among the non-responders is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: as for outcome 34
Measure: Mean (Standard Error); unit: Voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 12 | 12
Voxels | -465.5 (273.77) | -898.5 (554.98)

36. Secondary Outcome: Number of Contiguous Activated Voxels Meeting Predefined Threshold in the Thalamus on fMRI by 2-Back Working Memory Test-Change From Baseline; Subgroup-Non Responders in 2 Back Memory Test
Description: This is a subgroup analysis of non-responders on the 2-back working memory test for the number of voxels meeting the predefined threshold (voxels that differ significantly from reference wave form) on functional magnetic resonance imaging (fMRI). A non-responder in the 2-back working memory test was defined as a patient showing a response latency of 713 ms or greater at endpoint. The change from Baseline to Endpoint in the number of activated voxels in the thalamus for each treatment group among the non-responders is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: as for outcome 34
Measure: Mean (Standard Error); unit: Voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 12 | 12
Voxels | -893.1 (545.48) | -1408.3 (795.57)

37. Secondary Outcome: Change From Baseline to Endpoint in the BOLD Signal Intensity in the Dorsolateral Prefrontal Cortex (DLPFC) at Resting State
Description: At resting state, this is an analysis of the change from Baseline to Endpoint in the blood oxygen level dependent (BOLD) signal intensity in the dorsolateral prefrontal cortex (DLPFC).
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one observation after baseline
Measure: Median (Full Range); unit: BOLD signal intensity
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 17 | 16
BOLD signal intensity | 5.556 (57.6441) [-40.0 to 971.429] | 3.755 (5.0906) [-39.855 to 33.333]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.7053, Wilcoxon (Mann-Whitney); Median Difference (Net) = 4.841, 95% CI 2-sided [-27.778 to 19.313]

38. Secondary Outcome: Change From Baseline to Endpoint in the BOLD Signal Intensity in the Anterior Cingulate Cortex (ACC) at Resting State
Description: At resting state, this is an analysis of the change from Baseline to Endpoint in the blood oxygen level dependent signal (BOLD) intensity in the anterior cingulate cortex (ACC).
Time Frame: Baseline and Endpoint (Week 2 or last observation after Baseline)
Population: Full Analysis Set defined as subjects who had at least one observation after baseline
Measure: Median (Full Range); unit: BOLD signal intensity
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 17 | 16
BOLD signal intensity | 2.778 (9.6476) [-100.0 to 85.714] | 0.0 (7.2850) [-45.714 to 75.0]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.5163, Wilcoxon (Mann-Whitney); Median Difference (Net) = 4.792, 95% CI 2-sided [-30.631 to 16.190]

39. Secondary Outcome: Change From Baseline in the BOLD Signal Intensity in the Posterior Parietal Cortex (PPC) at Resting State
Description: At resting state, this is an analysis of the change from Baseline to Endpoint in the blood oxygen level dependent (BOLD) signal intensity in the posterior parietal cortex (PPC).
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who have had at least one observation after Baseline
Measure: Median (Full Range); unit: BOLD signal intensity
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 17 | 16
BOLD signal intensity | 2.667 (8.9840) [-25.0 to 144.444] | 2.479 (3.3927) [-32.283 to 18.831]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.8711, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0.108, 95% CI 2-sided [-14.341 to 5.498]

40. Secondary Outcome: Change From Baseline to Endpoint in the BOLD Signal Intensity in the Thalamus at Resting State
Description: At resting state, this is an analysis of the change from Baseline to Endpoint in the blood oxygen level dependent (BOLD) signal intensity in the thalamus.
Time Frame: Baseline and Endpoint (Week 2 or last observation after Baseline)
Population: Full Analysis Set defined as subjects who have had at least one observation after Baseline
Measure: Median (Full Range); unit: BOLD signal intensity
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 17 | 16
BOLD signal intensity | 5.128 (32.2812) [-30.769 to 544.444] | 1.429 (3.9156) [-29.204 to 22.222]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.1825, Wilcoxon (Mann-Whitney); Median Difference (Net) = 13.855, 95% CI [-15.357 to 25.714]

41. Secondary Outcome: Change From Baseline to Endpoint in the Number of Voxels Meeting Predefined Threshold in the Dorsolateral Prefrontal Cortex (DLPFC) at Resting State
Description: At resting state, this is an analysis of the change from Baseline to Endpoint in the number of contiguous activated voxels (voxels that differ significantly from reference wave form) on functional magnetic resonance imaging (fMRI) in the dorsolateral prefrontal cortex.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects who had at least one observation after Baseline
Measure: Median (Full Range); unit: Voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 17 | 16
Voxels | 941.5 (1613.73) [-12443.0 to 11600.0] | -174.5 (1418.92) [-9388.5 to 12014.0]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.9282, Wilcoxon (Mann-Whitney); Median Difference (Net) = -323.5, 95% CI 2-sided [-9311.0 to 2375.5]

42. Secondary Outcome: Change From Baseline to Endpoint in the Number of Voxels Meeting Predefined Threshold in Anterior Cingulate Cortex (ACC) at Resting State
Description: At resting state, this is an analysis of the change from Baseline to Endpoint in the number of contiguous activated voxels meeting pre-defined threshold (voxels that differ significantly from reference wave form) on functional magnetic resonance imaging (fMRI) in the anterior cingulate cortex (ACC).
Time Frame: Baseline and Endpoint (Week 2 or last observation after Baseline)
Population: Full Analysis Set defined as subjects with at least one observation after Baseline
Measure: Median (Full Range); unit: Voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 17 | 16
Voxels | -27.5 (197.41) [-1969.0 to 1229.5] | -54.0 (231.69) [-883.0 to 2750.0]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 1.0000, Wilcoxon (Mann-Whitney); Median Difference (Net) = 1.0, 95% CI 2-sided [-1069.0 to 426.0]

43. Secondary Outcome: Change From Baseline to Endpoint in the Number of Voxels Meeting Predefined Threshold in Posterior Parietal Cortex (PPC) at Resting State
Description: At resting state, this is an analysis of the change from Baseline to Endpoint in the number of activated voxels meeting predefined threshold (voxels that differ significantly from reference wave form) on functional magnetic resonance imaging (fMRI) in the posterior parietal cortex (PPC).
Time Frame: Baseline and Endpoint (Week 2 or last observation after Baseline)
Population: Full Analysis Set defined as subjects with at least one observation after Baseline
Measure: Median (Full Range); unit: Voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 17 | 16
Voxels | 22.0 (517.56) [-4602.0 to 759.0] | 104.3 (382.49) [-1994.5 to 1747.0]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.5284, Wilcoxon (Mann-Whitney); Median Difference (Net) = -82.8, 95% CI 2-sided [-788.0 to 165.5]

44. Secondary Outcome: Change From Baseline to Endpoint in the Number of Voxels Meeting Predefined Threshold in the Thalamus at Resting State
Description: At resting state, this is an analysis of the change from Baseline to Endpoint in the number of activated voxels meeting predefined threshold (voxels that differ significantly from reference wave form) on functional magnetic resonance imaging (fMRI) in the thalamus.
Time Frame: Baseline and Endpoint (Week 2 or last observation after baseline)
Population: Full Analysis Set defined as subjects with at least one observation after Baseline
Measure: Median (Full Range); unit: Voxels
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 17 | 16
Voxels | -621.0 (517.64) [-5251.0 to 3171.5] | -883.8 (689.30) [-5876.0 to 5806.0]
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.8997, Wilcoxon (Mann-Whitney); Median Difference (Net) = -145.8, 95% CI 2-sided [-3151.0 to 1006.5]

45. Secondary Outcome: Change From Baseline to Endpoint (2 Weeks or Last Observation After Baseline) in the Mean Response Latency in the Psychomotor Vigilance-Like Test
Description: During anatomic scanning (and prior to functional runs when anatomic scanning was not performed), a modified continuous 10 minute attention task ("Psychomotor Vigilance Test [PVT]-like task," nearly identical to the PVT but for absence of performance feedback) was run to obtain a measure of vigilance in the scanner-in this instance, the "+" symbol appeared at random (mean inter trial interval of 5 seconds, range 2 - 10 seconds) but disappeared when subject pressed a button. Subject performance speed was measured. Change in subject performance speed from Baseline to Endpoint is presented.
Time Frame: Baseline and Endpoint (Week 2 or last observation after Baseline)
Population: Full Analysis Set defined as subjects who had at least one observation after Baseline
Measure: Least Squares Mean (Standard Error); unit: milliseconds (ms)
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 15 | 15
milliseconds (ms) | -31.9 (13.41) | -6.8 (13.16)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p = 0.1305, ANCOVA; Mean Difference (Net) = -25.1, 95% CI 2-sided [-58.2 to 8.0]

ADVERSE EVENTS:
Time Frame: 2 Weeks
Arm/Group | Armodafinil (200 mg/Day) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 13/21 | 3/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil (200 mg/Day) (N=21) | Placebo (N=19)
Abdominal Pain upper (Gastrointestinal disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Bruxism (Psychiatric disorders) | 1 | 0
Cardiac murmur (Investigations) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1
Energy increased (General disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 1
Heart rate increased (Investigations) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Irritability (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pollakuria (Renal and urinary disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other